CLINICAL TRIAL: NCT05295082
Title: Accuracy of Trephination-based Versus Drilling-based Guided Dental Implant Placement: A Randomized Clinical Study
Brief Title: Accuracy of Trephination-based Versus Drilling-based Guided Dental Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Ramadan (Other)
Responsible Party: Sponsor-Investigator, Mohammed Ramadan, Principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecIM012225
Record Dates: First submitted 2022-03-03; First posted 2022-03-24 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Single Tooth Lost; Partially Edentulous Maxilla
Keywords: guided implant; surgical guide; dental implant; dental trephination; guided trephination

STUDY DESIGN:
Intervention Model Description: guided dental implant placement through guided trephine-based implant site preparation
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor is not involved in the study. he doesn't know the type of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided trephination-based protocol (Experimental): The drilling process will be performed by guided trephination protocol.
  * An appropriate trephine drill (Helmut Zepf Medizintechnik GmbH, Germany) will be used to create an initial osteotomy.
  * The guide will be removed, and the depth and angulation of this initial osteotomy will be evaluated.
  * The final drill of the chosen implant system will be used to complete the osteotomy.
  * The implant (NeoBiotech Implant System, Neobiotech Co. Ltd. Korea) then will be placed freehand in a conventional manner.
  Interventions: Procedure: guided trephination-based drilling protocol
- guided conventional drilling-based protocol (Active Comparator): The drilling process will be performed by a guided conventional drilling protocol.
  * Drilling (Neo NaviGuide System - Neobiotech Co. Ltd. Korea) will be performed throughout the guiding sleeve from the first drill to the final drill.
  * The guide will be removed.
  * The implant (NeoBiotech Implant System, Neobiotech Co. Ltd. Korea) then will be placed freehand in a conventional manner.
  Interventions: Procedure: guided Conventional drilling-based protocol

INTERVENTIONS:
Procedure: guided trephination-based drilling protocol — the implant site preparation in this group will be done by guided trephination protocol which uses the surgical guide to trephine the implant site then remove the guide and continue the drilling in a freehand manner
  Arms: guided trephination-based protocol
Procedure: guided Conventional drilling-based protocol — the implant site preparation in this group will be done by a guided conventional drilling protocol which uses the surgical guide to guide the sequential drills up to the final drill
  Arms: guided conventional drilling-based protocol

SUMMARY:
This study will be initiated to compare the accuracy of implant placement using the guided trephination drilling protocol and the guided conventional drilling protocol.

DETAILED DESCRIPTION:
This study will be conducted to compare the accuracy of implant placement using the guided trephination drilling protocol and the guided conventional drilling protocol.

the patients with a single missing tooth will be assigned to one group ( trephination drilling / conventional drilling ).the preoperative virtual planning and fabrication of a surgical guide will be made for each patient. after implant placement according to each group, postoperative (CBCT ) will be performed to compare the virtual implant position and the actual implant position.

ELIGIBILITY:
Inclusion Criteria:

1. Single missing maxillary premolar or molar tooth.
2. Both genders aged from 20-50 years.
3. Patients should be systematically free from any disease as according to Cornell Medical Index-Health Questionnaire. (Pendleton et al,.2004)
4. Mesio-distal space ≥ 7 mm.
5. Bone width in bucco-lingual direction ≥ 6 mm.
6. Uniform alveolar ridge with no undercuts.
7. Present mesial and distal sound neighboring teeth.
8. At least 4 natural remaining teeth on the same arch.
9. Mouth opening at least 30 mm.

Exclusion Criteria:

1) Pregnant and lactating females. 2) Smokers. 3) Poor oral hygiene. 4) Vulnerable groups of patients' e.g. (handicapped patients).

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Horizontal deviation at apex of the implant. | immediately after the intervention
  measure the Horizontal deviation at apex of the implant between the virtual planning position and the actual implant position
•Horizontal deviation at implant shoulder. | immediately after the intervention
  measure the Horizontal deviation at the implant shoulder between the virtual planning position and the actual implant position
Angular deviation. | immediately after the intervention
  measure the Angular deviation of the implant between the virtual planning position and the actual implant position

SECONDARY OUTCOMES:
The duration of the surgery | during the surgery
  measure the time of the surgery from the first drill to the implant placement
Satisfaction assessed by the Visual Analogue Scale | immediately after the intervention
  measure the patient satisfaction score on terms of pain and discomfort from 1 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the data that will be shared is the CBCT, virtual planning

REFERENCES:
- [Result] Suriyan N, Sarinnaphakorn L, Deeb GR, Bencharit S. Trephination-based, guided surgical implant placement: A clinical study. J Prosthet Dent. 2019 Mar;121(3):411-416. doi: 10.1016/j.prosdent.2018.06.004. Epub 2018 Nov 30. PMID 30503150
- [Result] Van Assche N, Vercruyssen M, Coucke W, Teughels W, Jacobs R, Quirynen M. Accuracy of computer-aided implant placement. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:112-23. doi: 10.1111/j.1600-0501.2012.02552.x. PMID 23062136
- [Result] Cassetta M, Stefanelli LV, Giansanti M, Di Mambro A, Calasso S. Accuracy of a computer-aided implant surgical technique. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):317-25. doi: 10.11607/prd.1019. PMID 23593625